CLINICAL TRIAL: NCT06790654
Title: Text-based Motivational Interviewing Intervention to Promote Exclusive Breastfeeding Rates
Acronym: Text-MI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-465
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breastfeeding Rate; Breastfeeding Self-Efficacy
Keywords: breastfeeding; motivational interviewing
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Motivational interviewing (Experimental): All participants will receive the intervention which consists of 6 weeks of text-based motivational interviewing targeted at addressing barriers to exclusive breastfeeding.
  Interventions: Behavioral: Text-message based motivational interviewing

INTERVENTIONS:
Behavioral: Text-message based motivational interviewing — Participants will receive weekly text messages during the pilot study period, initiated and managed by MItrained interviewers. Each text message exchange will begin with a short, MI-consistent prompt developed with input from focus groups of mothers who have previously breastfed. These prompts will address common breastfeeding barriers. Following the initial prompt, MI-trained trainers will engage with participants through text exchanges that utilize the core MI OARS skills (open-ended questions, affirmations, reflections, or summaries) to facilitate change talk.

SUMMARY:
The goal of this clinical trial is to evaluate whether a text-based motivational interviewing (MI) intervention can increase exclusive breastfeeding rates and breastfeeding self-efficacy in mothers of healthy full-term infants. This study focuses on addressing breastfeeding barriers, particularly among mothers in underserved and rural populations.

The main questions it aims to answer are:

* Does a text-based MI intervention improve exclusive breastfeeding rates at two, four, and six weeks postpartum?
* Does the intervention increase maternal breastfeeding self-efficacy during the same period?

Researchers will compare the outcomes of mothers receiving the text-based MI intervention to standard breastfeeding support to assess its feasibility, acceptability, and initial effectiveness.

Participants will:

* Receive weekly personalized motivational text messages for six weeks postpartum.
* Engage in interactive exchanges with MI-trained interviewers addressing breastfeeding challenges.
* Complete surveys at baseline, mid-intervention, and post-intervention to assess breastfeeding behaviors and self-efficacy.

DETAILED DESCRIPTION:
Overview This pilot study will develop and evaluate the feasibility and acceptability of a text-based motivational interviewing intervention to increase breastfeeding rates. Mother-infant dyads will be recruited from the University of Mississippi Medical Center full-term nursery. Tailored text messages will address breastfeeding barriers, informed by focus groups and an expert panel. We will assess adherence, satisfaction, and fidelity and explore initial changes in breastfeeding self-efficacy and breastfeeding rates at two, four, and six weeks to inform the development of a clinical trial.

Aim 1: To develop a text-based motivational interviewing (MI) intervention and procedures for delivery.

We will use focus groups to gather qualitative data on breastfeeding barriers and integrate feedback from these groups and experts to tailor messages that reflect parent needs. We will recruit 6-8 mothers through Health Moms Health Babies (MSDH), MOM. M.E. via Mental Health Mississippi, La Leche League of Metro Jackson, MS Breastfeeding Coalition Facebook group, and the EversCare Clinic (via UMMC). We will facilitate 2-3 focus group sessions, each lasting approximately 1.5 to 2 hours, using a semi-structured interview guide to explore participants' experiences and challenges with breastfeeding. This qualitative analysis will aim to identify common barriers to exclusive breastfeeding that can be addressed through the MI protocol. The sessions will be recorded, transcribed, and analyzed qualitative data to identify and categorize themes related to barriers to exclusive breastfeeding.

Next, we will engage experts in motivational interviewing, lactation, and neonatology to ensure the messaging strategy is appropriate, evidence-based, and effectively addresses barriers to breastfeeding. We will employ the Delphi Technique, involving multiple rounds of anonymous questionnaires distributed to a panel of experts. Experts will provide feedback on the MI-based text messages in each round, which will be summarized and shared with the panel before the next round. The iterative nature of the Delphi Technique will help achieve consensus on the most effective and culturally sensitive messages for our intervention.

Procedures for Delivery

Platform Implementation (Twilio and REDCap). The delivery of the text messages will be implemented using Twilio, a messaging API, integrated with the HIPAA-compliant REDCap application. This integration will enable automated scheduling and delivery of personalized messages and reminders based on the MI protocol. Twilio will provide valuable metadata on response rates and engagement patterns. We will create and configure a Twilio account specifically for this study, setting up messaging services, acquiring necessary phone numbers, and ensuring compliance with HIPAA regulations. Twilio will be integrated with REDCap to manage participant data securely.

Developing Message Workflows. MI-trained interviewers will utilize the infrastructure set up in REDCap to guide their interactions, allowing for real-time adaptation of message content based on participant feedback. This approach ensures that the intervention remains dynamic and responsive to individual needs.

Training and Monitoring. Site P.I.s and study coordinators will receive training from a certified MI Network Trainer (MINT) on the MI principles and the specifics of the message bank content. This training will ensure that the intervention adheres to MI principles and is implemented consistently. Throughout the pilot, a sample of text exchanges will be monitored weekly to ensure fidelity to MI principles. Adjustments will be made as needed based on these reviews.

Aim 2: Evaluate the Feasibility and Acceptability of the 24-Week Text-Based MI Intervention We will pilot our intervention over six weeks with mother-infant dyads recruited from the University of Mississippi Medical Center's term baby nursery. Inclusion criteria include mothers with healthy-term infants, cell phone access, and intent to breastfeed. Exclusion criteria include age < 18, contraindications to breastfeeding, substance use, or multiple gestation.2 We aim to recruit 30 mothers. Participants will receive $75 as an incentive for their participation. Participants will follow the schedule of events shown in Table 1.

Intervention Plan Participants will receive weekly text messages during the pilot study period, initiated and managed by MI-trained interviewers. Each text message exchange will begin with a short, MI-consistent prompt developed with input from focus groups of mothers who have previously breastfed. These prompts will address common breastfeeding barriers. Following the initial prompt, MI-trained trainers will engage with participants through text exchanges that utilize the core MI OARS skills (open-ended questions, affirmations, reflections, or summaries) to facilitate change talk. Additional MI tools, such as change rulers, will be employed to support participants in setting goals for the upcoming week. Each exchange will be limited to five delivered text messages and five participant replies, ensuring focused and effective communication. All MI-trained trainers will undergo a comprehensive training program conducted by a certified MI Network Trainer (MINT). This program will include detailed sessions on the specific requirements of the text-based intervention, with a strong focus on practicing and refining MI techniques suitable for text messaging. Ongoing supervision will be provided throughout the study to ensure consistent application of MI principles and address any challenges that arise during the intervention.

Measures Feasibility. To assess feasibility, we will monitor several key indicators. Intervention adherence will be tracked by monitoring message delivery and participant engagement using system usage data. The number of messages successfully delivered, and the response rate to interactive messages will be recorded. Adherence rates will be calculated as the proportion of delivered messages to the total number of scheduled messages, and the engagement rate will be calculated based on participant interactions with the messages. Recruitment and retention rates will be monitored by tracking the number of participants recruited, enrolled, and retained throughout the study. Recruitment success will be measured by the proportion of eligible mothers who agree to participate. Retention will be assessed by the proportion of participants who complete the intervention. Recruitment and retention rates will be reported as percentages, and reasons for dropout will be documented and analyzed to identify potential barriers to retention.

Acceptability. To evaluate acceptability, we will gather both quantitative and qualitative data from participants. Participant satisfaction with the intervention will be assessed using surveys that include questions on the text messages' relevance, clarity, helpfulness, and overall satisfaction. The surveys will be administered at baseline, mid-intervention, and post-intervention. Survey responses will be analyzed using descriptive statistics to summarize participant satisfaction and identify areas for improvement. We will collect qualitative feedback through follow-up interviews or focus groups with a subset of participants at the end of the intervention. A semi-structured interview guide will be used to explore participants' perceptions of the intervention's strengths and weaknesses. Qualitative data will be transcribed and analyzed thematically to identify common themes and suggestions for refining the intervention.

Implementation Fidelity. Adherence to the intervention protocol will be verified by ensuring that the correct messages are sent at the scheduled times and that the platform functions as intended. This will involve regular checks and audits of the message delivery system. Protocol adherence will be reported as the proportion of messages sent on time, and any deviations from the protocol will be documented and analyzed. Comprehensive training sessions will be provided for the staff involved in delivering the intervention and conducting follow-up assessments. Training will cover the use of the text message platform, adherence to the intervention protocol, and techniques for collecting qualitative data. Regular supervision and meetings will be held to address any issues and ensure fidelity to the intervention protocol. Feedback from staff will be collected and used to improve training and supervision processes. A random sample of text message exchanges will be reviewed periodically by an MI expert. This expert, preferably a certified MI Network Trainer (MINT), will evaluate the exchanges for adherence to MI techniques and overall alignment with the intervention's goals. The expert will provide a detailed feedback report after each review, highlighting strengths and suggesting areas for improvement.

Aim 3: Explore Preliminary Changes in Breastfeeding Self-Efficacy and Exclusive Breastfeeding Rates

Aim 3 seeks to understand the intervention's impact on breastfeeding self-efficacy and exclusive breastfeeding rates over time. To do this, we will measure these outcomes at baseline, mid-intervention, and post-intervention using a survey instrument that includes the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) and measures of breastfeeding practices adapted from CDC's Infant Feeding Practices Study II.23,24These data points will be collected through REDCap surveys administered at the specified intervals. To analyze these data, we will employ mixed-effects models. Specifically, linear mixed models will be used to assess changes in breastfeeding self-efficacy, incorporating time as a fixed effect and allowing for random effects to capture individual variability. For exclusive breastfeeding rates, which are categorical, logistic mixed models will analyze the likelihood of exclusive breastfeeding across the study period, adjusting for potential confounders identified at baseline. We will also examine potential subgroup differences (e.g, age, partity, education level) to refine the randomization and stratification process. These results will provide preliminary estimates of the intervention's potential effectiveness and guide the design and sample size calculations for a future full-scale trial, ensuring it is appropriately designed and adequately powered to detect significant effects.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have given birth to a healthy full-term infant, intend to breastfeed, and possess a mobile device capable of receiving texts

Exclusion Criteria:

* Exclusion criteria include age < 18, contraindications to breastfeeding, substance use, or multiple gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Enrollment Number | End of study (six weeks)
  As a pilot measure of study feasibility, the final sample of participants will be compared against the target sample size of 30.
Retention | End of study (six weeks)
  Retention will be calculated as the percentage of participants who complete the study out of those enrolled.
Adherence | End of study (six weeks)
  Adherence (consistency of engagement with the text messages) will be measured as the share of interview sessions in which participants' respond to at least one motivational interviewing prompt.
Acceptability | End of study (6 weeks)
  Acceptability will be assessed using an measure of participant satisfaction with the program. This measure is a 5-item scale covering overall experience, clarity of text messages, helpfulness of guidance, influence on breastfeeding practices, and likelihood of recommending the program to others. Each item will be rated on a 5-point Likert scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Scores will be summed to produce a total satisfaction score, ranging from 5 to 25, with higher scores reflecting greater satisfaction.
Exclusive breastfeeding rates | Weeks 3 and 6 of the intervention.
  Exclusive breastfeeding status will be self-reported by participants.

SECONDARY OUTCOMES:
Mixed-breastfeeding rates | Weeks 3 and 6 of the intervention.
  Rates of breastfeeding with supplementation will be reported by participants.
Breastfeeding Self-Efficacy | Enrollment, week 3, and week 6.
  Breastfeeding self-efficacy will be measured using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF). the BSES-SF is a 14-item with each item rated on a 5-point Likert scale, ranging from 1(not at all confident) to 5(always confident). The items will be summed to produced a total ranging from 14 to 70 with higher scores representing greater self-efficacy.